CLINICAL TRIAL: NCT00962819
Title: Persistence of Humoral and Cellular Immune Responses Following Age-appropriate Vaccination With the MMR Vaccine
Brief Title: Measles, Mumps, and Rubella (MMR) Immunity in College Students
Status: Completed | Type: Observational
Sponsor: Sri Edupuganti, MD MPH (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Sri Edupuganti, MD MPH, Assistant Prfessor, Emory University
Organization: Emory University (Other)
Other Study IDs: IRB00007373
Record Dates: First submitted 2008-05-19; First posted 2009-08-20 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Measles; Mumps; Rubella
Keywords: Mumps; Immunity; Vaccine; Mumps antibodies; Mumps immunity
MeSH Terms: conditions — Measles; Mumps; Rubella | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cross-sectional: College-aged students who were immunized with MMR.
  Interventions: Biological: MMR vaccine

INTERVENTIONS:
Biological: MMR vaccine — People with no antibodies to either mumps, measles and rubella will be offered the MMR vaccine (they may choose to or choose not to receive the MMR vaccine)
  Other Names: No other names

SUMMARY:
This study will lay the foundation for determining the underlying reasons for lack of immunity to mumps that led to the 2006 mumps outbreak on college campuses in the Mid West, and it will assess the potential for similar outbreaks of measles and rubella. A total of 70 to 80 college students (age 18 to 22) on the Emory campus (or nearby college campuses or the community) will be assessed for antibodies to measles, mumps or rubella by drawing a one-time blood sample. Their medical records will be verified for documentation of immunization with MMR vaccine prior to enrollment in the study. If a study volunteer is found to not have MMR immunity, they will be offered an MMR-II vaccine. For this group, additional blood specimens will be obtained.

DETAILED DESCRIPTION:
No additional description needed.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willing to provide an informed consent
* Documented receipt of MMR-II vaccination in childhood
* Not pregnant

Exclusion Criteria

* No history of HIV infection.
* Immunocompromised health status due to HIV infection, cancer, diabetes, liver, lung or kidney diseases, autoimmune diseases, history of splenectomy.
* Use of immunosuppressive medications within last 2 to 3 months (oral or parenteral corticosteroids or cytotoxic medications)
* Medical conditions that require the use of immunosuppressive medications
* Received blood or blood products within the last 30 days
* Any vaccines received in the last 30 days

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects for this study will be 18-22 year olds recruited from Emory University's student population who have received two age-appropriate doses of the MMR-II vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Levels of mumps antibody and levels of memory B and T cell responses | Day 1 for all participants except for those who receive MMR vaccine, there will be additional outcome measures on Day 0, 7, 14 and 28 post-vaccination.
  Cross sectional measurement of antibodies to mumps. measles or rubella

SECONDARY OUTCOMES:
Determine proportion of college-aged students who are seronegative for mumps | outcome measurement on Day 1
  Cross-sectional measurement of antibodies to mumps, measles and rubella

CONTACTS AND LOCATIONS:
Overall Officials: Srilatha Edupuganti, MD, Principal Investigator — Emory University
Locations (1):
- The Hope Clinic of the Emory Vaccine Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dayan GH, Quinlisk MP, Parker AA, Barskey AE, Harris ML, Schwartz JM, Hunt K, Finley CG, Leschinsky DP, O'Keefe AL, Clayton J, Kightlinger LK, Dietle EG, Berg J, Kenyon CL, Goldstein ST, Stokley SK, Redd SB, Rota PA, Rota J, Bi D, Roush SW, Bridges CB, Santibanez TA, Parashar U, Bellini WJ, Seward JF. Recent resurgence of mumps in the United States. N Engl J Med. 2008 Apr 10;358(15):1580-9. doi: 10.1056/NEJMoa0706589. PMID 18403766
- [Result] Rasheed MAU, Hickman CJ, McGrew M, Sowers SB, Mercader S, Hopkins A, Grimes V, Yu T, Wrammert J, Mulligan MJ, Bellini WJ, Rota PA, Orenstein WA, Ahmed R, Edupuganti S. Decreased humoral immunity to mumps in young adults immunized with MMR vaccine in childhood. Proc Natl Acad Sci U S A. 2019 Sep 17;116(38):19071-19076. doi: 10.1073/pnas.1905570116. Epub 2019 Sep 3. PMID 31481612
- See also: website for vaccine research clinic — http://www.medicine.emory.edu/id/hopeclinic/